CLINICAL TRIAL: NCT06997159
Title: A Randomized, Multicentre, Observer-blind Phase II Study to Evaluate the Efficacy, Safety and Pharmacokinetics (PK) of Two LXE408 Regimens and Miltefosine as an Active Control in Patients With Localized Cutaneous Leishmaniasis in the Region of the Americas (AMR).
Brief Title: A Clinical Trial to Investigate Efficacy, Safety and Pharmacokinetics (PK) of Two LXE408 Oral Regimens and Oral Miltefosine as Active Control in Participants Aged ≥ 18 Years Old With Localized Cutaneous Leishmaniasis in the Region of the Americas (AMR).
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DNDi-LXE408-03-CL; CLXE408C12201R (Other: Novartis)
Record Dates: First submitted 2025-05-13; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Localized Cutaneous Leishmaniasis
Keywords: Localized Cutaneous Leishmaniasis
MeSH Terms: interventions — LXE408; miltefosine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants and investigators are partially blinded: they will be blinded for the two investigational LXE408 arms, which will reduce bias in the clinical assessment of safety and efficacy. However, both participants and investigators will be aware whether they are assigned to the investigational arms or to the miltefosine arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- LXE408 BID for 14 days (Experimental): LXE408 BID for 14 days followed by placebo BID for 14 days.
  Interventions: Drug: LXE408; Drug: Placebo to LXE408
- LXE408 BID for 28 days (Experimental)
  Interventions: Drug: LXE408
- Miltefosine 50 mg PO TID for 28 days (Active Comparator)
  Interventions: Drug: Miltefosine 50 MG Oral Capsule [Impavido]

INTERVENTIONS:
Drug: LXE408 — LXE408 film-coated tablets.
  Arms: LXE408 BID for 14 days; LXE408 BID for 28 days
Drug: Miltefosine 50 MG Oral Capsule [Impavido] — Each capsule contains 50 mg miltefosine in an opaque, red, hard gelatin capsule. Capsules are supplied in packs of 56 capsules sealed in 8 aluminum blister stripes, each containing 7 capsules.
  Arms: Miltefosine 50 mg PO TID for 28 days
Drug: Placebo to LXE408 — Film-coated tablets.
  Arms: LXE408 BID for 14 days

SUMMARY:
The purpose of this clinical trial is to measure efficacy, safety and pharmacokinetics (PK) of two LXE408 oral regimens and oral miltefosine tablets as active control in localized cutaneous leishmaniasis in the region of the Americas (AMR), and assess its suitability for use in monotherapy for the treatment of patients with cutaneous leishmaniasis (CL).

DETAILED DESCRIPTION:
Participants who met all inclusion criteria and none of the exclusion criteria will be randomized to the study will be allocated to one of three arms in a 2:2:1 ratio.

* Arm 1: LXE408 BID for 14 days followed by placebo BID for 14 days
* Arm 2: LXE408 BID for 28 days
* Arm 3: Miltefosine 50 mg PO TID for 28 days orally

Each arm will consist of a screening period of up to 15 days, a 28-day treatment period, and a follow-up period from Day 29 to Day 180. During the treatment period, all participants will return to the sites at Days 1, 8, 15, 22 and 29 (+/- 2 days). During the follow-up period they will return for the Day 63 (+/- 7 days), Day 90 (+/- 7 days) and Day 180 (+/- 14 days) visits. If at D90 participants present a re-epithelization of the ulcer(s) more or equal to 75% but less than 100%, they will be asked to return at D105 for a late responder assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be aged ≥18 years old and weighing > 50kg
2. Participant with first episode of CL fulfilling the following characteristics:

   * ≤ 6 lesions
   * At least one lesion of > 50 mm2 of area
   * a history of CL of no longer than 6 months
3. a diagnosis of CL confirmed by at least one of the following methods:

   * microscopic identification of amastigotes in stained lesion tissue, or
   * demonstration of Leishmania by PCR, or
   * positive culture for promastigotes
4. In the opinion of the investigator, the participant is capable of understanding and complying with the protocol, including visits up to 6 months after study start.
5. Written informed consent must be obtained before any study protocol specific assessment is performed other than procedures performed as part of standard of care.

Participants must be able to give written informed consent.

Exclusion Criteria:

1. Female with a positive blood pregnancy test at screening or who is breastfeeding, lactating or women of childbearing potential (defined as women physiologically capable of becoming pregnant) who does not agree to use two methods of contraception, one barrier method and one highly effective method. In Brazil: for 30 days prior to the treatment onset and up to D180 visit. In Panama: during treatment period up to D180 visit.
2. Sexually active male, including those post-vasectomy, unwilling to use a condom during intercourse with female partner while taking the investigational drug and for 5 days, after stopping the investigational drug.
3. Has diagnosis or suspected diagnosis of mucocutaneous, disseminated or diffuse leishmaniasis based on physical exam.
4. Current clinically significant medical problems (e.g., cardiac, renal, hepatic, pancreatic diseases, current cutaneous conditions that may interfere with CL evolution or healing, past and current ocular disorders, especially keratitis, uveitis, scleritis), including any immunocompromising condition (such as having a known diagnosis for HIV, transplanted patients, those in treatment for auto immune diseases, patients receiving immunosuppressant, immunobiological or antineoplastic treatments).
5. History of lymphoproliferative disease or any known malignancy or history of malignancy of any organ system within the past 5 years (except for basal cell carcinoma or actinic keratosis that have been treated with no evidence of recurrence in the past 3 months, carcinoma in situ of the cervix or non-invasive malignant colon polyps that have been removed).
6. Participants newly diagnosed with HIV infection on the basis of the trial screening testing or other recent testing (< 6 months) are excluded. Participants with documented stable HIV infection are allowed to participate in the study. Stable HIV infection is defined as: clinically stable with no signs or symptoms of advanced HIV infection and taking their current anti-retroviral therapy for ≥ 6 months with an undetectable viral load for ≥ 6 months. Participants taking anti-retroviral therapy prohibited in Section 6.9.4 are excluded.
7. Participants with active infectious conditions, such as tuberculosis, or history or active hepatitis B virus (HBV) infection or hepatitis C virus (HCV) infection are excluded. Active HBV is defined as a positive HBV surface antigen (HBsAg) test, or if standard local practice, a positive HBV core antigen test and all participants with a positive HBV core antibody screening test must have HBsAg measured. Active HCV is defined as having detectable HCV RNA and all participants with a positive HCV antibody test at screening must have HCV RNA measured. Participants taking therapy for HBV or HCV are excluded.
8. ECG abnormalities, either historic (no longer present) or current which, in the view of the investigator, indicate a significant risk to study participation. These include, but are not limited to, the following:

   * Clinically significant cardiac arrhythmias (e.g., sustained ventricular tachycardia and clinically significant second- or third-degree AV block without a pacemaker).
   * QTcF ≥450 ms.
   * History of familial long QT syndrome or known family history of Torsades de Pointes.
   * Resting heart rate (physical exam or 12 lead ECG) <60 bpm.
9. Participants who are receiving or have received antileishmanial medication, or prohibited medication or any medication that might interfere with the therapeutic response or cause harmful interactions with study medications, as defined in concomitant treatments in Section 6.9.4.
10. Has laboratory values at screening as follows:

    Serum creatinine: ≥1.5 times ULN*, ALT, AST, GGT, ALP: >1.5 times above upper normal level*. Total bilirubin > 1.5 times ULN* amylase or lipase > 1.5 times ULN*

    *Normal ranges obtained from local laboratory.
11. Known history of addiction/ alcohol abuse.
12. Hypersensitivity to miltefosine or any study medication excipients.
13. Participants with Sjogren-Larsson Syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-11-16 (Estimated); Primary Completion 2027-07-10 (Estimated); Study Completion 2027-07-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who achieved Cure at Day 180 | 180 days
  Cure at Day 180 (D180) is defined as:
  * 100% re-epithelialization of ulcerated lesions (if any) or flattening and/or no signs of induration of non-ulcerated lesions (if any) up to and at D90 and,
  * no relapse by D180, and
  * no rescue therapy up to D180
  * no death, regardless of cause, up to D180

SECONDARY OUTCOMES:
Proportion of participants with treatment-emergent adverse events (TEAEs) and SAEs | 180 days
Proportion of participants with • Abnormalities from physical exam, vital signs, ECGs and safety laboratory assessments | 180 days
Proportion of participants who achieved Cure at Day 90 | 90 days
  Cure at Day 90 (D90) is defined as:
  * 100% re-epithelization of ulcerated lesions (if any) or flattening and/or no signs of induration of non-ulcerated lesions (if any) at D90;
  * no rescue therapy up to D90.
  * No-death regardless of cause up to D90.
Pharmacokinetics (PK) of LXE408 - Cmax | Day 1, Day 8 and Day 15
  Maximum plasma concentration
Pharmacokinetics (PK) of LXE408 - Tmax | Day 1, Day 8 and Day 15
  Time to maximum plasma concentration
Pharmacokinetics (PK) of LXE408 - AUCtau | Day 1, Day 8 and Day 15
  Area under plasma concentration-time curve over dosing interval
Proportion of participants who achieved cure in different species of Leishmania for participants treated with LXE408 and miltefosine | Day 90, Day 180

CONTACTS AND LOCATIONS:
Locations (5):
- Brazil (4):
  - Foundation of Tropical Medicine Dr. Heitor Vieira Dourado, Manaus, Amazonas
  - Federal University of Maranhão, São Luís, Maranhão
  - Julio Muller University Hospital/ Federal University of Mato Grosso, Cuiabá, Mato Grosso
  - René Rachou Institute /Oswaldo Cruz Foundation- FIOCRUZ MINAS, Belo Horizonte, Minas Gerais
- Instituto Conmemorativo Gorgas de Estudios de la Salud, Panama City, Panama

IPD SHARING:
Plan to Share IPD: Yes